CLINICAL TRIAL: NCT02461173
Title: Comparison Between Stimulated Intrauterine Insemination Cycles and Unstimulated Intrauterine Insemination Cycles in Couples With Unexplained Infertility
Brief Title: Stimulated Intrauterine Insemination Cycles and Unstimulated Intrauterine Insemination Cycles in Couples With Unexplained Infertility
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sub 10
Record Dates: First submitted 2015-05-29; First posted 2015-06-03 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — hMG-IBSA; Ovulation Detection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stimulated IUI (Active Comparator): On the 3rd day of menstruation women in group 1 will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins starting from the 3nd day of menstruation. On day 8 the ultrasound will be repeated and serum E2 will be measured, hMG dose will be adjusted and continued and the frequency of ultrasound scans will be individualized. HMG will be stopped when at least 2 follicles measuring 18 mm are associated with serum E2 of 500-3000 Pg/mL, this was followed by the administration of 10000 IU of human chorionic gonadotropin
  Interventions: Drug: Merional; Procedure: IUI; Drug: Choriomon; Device: shepherd catheter
- Unstimulated IUI (Active Comparator): Women in group 2 will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit. IUI will be performed on the day after the surge in urinary excretion of luteinizing hormone.
  Interventions: Procedure: IUI; Procedure: Ovulation detection; Device: shepherd catheter
- Control group (Active Comparator): Women will be asked to test their urine for luteinizing hormone by the same method as group 2. They will be asked to have an intercourse on the day after the surge in urinary excretion of luteinizing hormone and this will be repeated for 12 months.
  Interventions: Procedure: Ovulation detection

INTERVENTIONS:
Drug: Merional — On the 3rd day of menstruation women will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins (hMG, Merional ®, IBSA, Lugano, Switzerland) starting from the 3nd day of menstruation.
  Arms: Stimulated IUI
Procedure: IUI — Semen will be processed and drawn into a shepherd catheter attached to a 1 mL syringe and injected into the uterus
  Arms: Stimulated IUI; Unstimulated IUI
Procedure: Ovulation detection — Women will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit
  Arms: Control group; Unstimulated IUI
Drug: Choriomon — Administration of 10000 IU of human chorionic gonadotropin (hCG; Choriomon®, IBSA) when at least 2 follicles measuring 18 mm are observed during vaginal ultrasound and is associated with serum E2 of 500-3000 Pg/mL
  Arms: Stimulated IUI
Device: shepherd catheter
  Arms: Stimulated IUI; Unstimulated IUI

SUMMARY:
Four hundred and fifty women with unexplained infertility will be divided into 3 equal groups using computer generated random numbers: Group 1 will have up to 4 stimulated IUI cycles, group 2 will have up to 4 unstimulated cycles, women who do not become pregnant after the 4 cycles in groups 1 and 2 will be advised to have regular intercourse at the expected time of ovulation. Group 3 will be the control group will be advised to have regular sexual intercourse at the time of ovulation for 6 months

DETAILED DESCRIPTION:
Unexplained infertility is a common diagnosis encountered in the subfertility clinic; about 15-30% of infertile couples will be diagnosed as having unexplained infertility. Couples are usually diagnosed as having unexplained infertility if the woman has ovulatory cycles, patent tubes and the spouse has a normal semen analysis according to the world health organisation criteria.

In the absence of an organic abnormality or a clear functional defect, couples with unexplained infertility have been subjected to several empirical treatments including intra-uterine insemination (IUI). The application of ovarian stimulation in IUI is advocated, even if the woman has ovulatory cycles, to improve the pregnancy rates with IUI. However, the application of ovarian stimulation has two main drawbacks: The increased chances of a multiple pregnancy and ovarian hyperstimulation syndrome. To avoid these complications unstimulated IUI cycles have been investigated. The objective of the study is to evaluate the role of stimulated and unstimulated IUI cycles in the management of unexplained infertility.

The study will be conducted in Cairo university hospitals and BeniSuef University hospitals All patients with unexplained infertility attending both sites will be invited to participate in the study. The study will be explained and only couples who sign written consents will be included in the study.

Four hundred and fifty women with unexplained infertility will be divided into 3 equal groups using computer generated random numbers: Group 1 will have up to 4 stimulated IUI cycles, group 2 will have up to 4 unstimulated cycles, women who do not become pregnant after the 4 cycles in groups 1 and 2 will be advised to have regular intercourse at the expected time of ovulation. Group 3 will be the control group will be advised to have regular sexual intercourse at the time of ovulation for 6 months On the 3rd day of menstruation group 1 will have a vaginal ultrasound and will receive daily intramuscular 150 IU of human menopausal gonadotropins (hMG, Merional ®, IBSA, Lugano, Switzerland) starting from the 3nd day of menstruation. On day 8 the ultrasound will be repeated and serum E2 will be measured, hMG dose will be adjusted and continued and the frequency of ultrasound scans will be individualized. HMG will be stopped when at least 2 follicles measuring 18 mm are associated with serum E2 of 500-3000 Pg/mL, this was followed by the administration of 10000 IU of human chorionic gonadotropin (hCG; Choriomon®, IBSA) Women in group 2 will be asked to test their morning urine specimen for luteinizing hormone daily starting 4 days before the expected day of ovulation. This will be done using a qualitative kit. Intrauterine insemination will be performed on the day after the surge in urinary excretion of luteinizing hormone.

Women in group 3 will be asked to test their urine for luteinizing hormone by the same method as group 2. They will be asked to have an intercourse on the day after the surge in urinary excretion of luteinizing hormone and this will be repeated for 12 months.

Semen specimens for groups 1 and 2 will be evaluated and prepared for IUI within one hour after collection. Semen will be diluted 1:2 (vol/vol) with HEPES-buffered Ham's F10 medium containing 1.5 percent serum albumin. After centrifugation for 10 minutes, the pellets will be resuspended and combined in 3 ml of the medium.

The sperm suspension will be centrifuged for 10 minutes, and the pellet was resuspended in 0.35 ml of medium. Approximately 0.05 ml will be used to determine the concentration and motility of sperms. The remaining sample will be drawn into a shepherd catheter attached to a 1 mL syringe and injected into the uterus.

The procedure will be repeated for up to 4 months in groups 1 and 2, if pregnancy does not occur. Women who do not conceive after the 4 trials will be asked to check their urine for luteinizing hormone using the ovulation detection kits and have an intercourse on the day following the luteinizing hormone surge. This will be repeated for 8 months.

The pregnancy rates of the 3 groups will be compared after the 4 months and after one year.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility

Exclusion Criteria:

* Known allergy to FSH
* Diabetes, hypertension, known cardiac, renal or liver disease.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ongoing pregnancy | 12 weeks after IUI or timed sexual intercourse
  confirmation of a viable pregnancy by detecting fetal heart beat during abdominal ultrasound examination

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Brandes M, Hamilton CJ, van der Steen JO, de Bruin JP, Bots RS, Nelen WL, Kremer JA. Unexplained infertility: overall ongoing pregnancy rate and mode of conception. Hum Reprod. 2011 Feb;26(2):360-8. doi: 10.1093/humrep/deq349. Epub 2010 Dec 16. PMID 21163857
- [Background] Cooper TG, Noonan E, von Eckardstein S, Auger J, Baker HW, Behre HM, Haugen TB, Kruger T, Wang C, Mbizvo MT, Vogelsong KM. World Health Organization reference values for human semen characteristics. Hum Reprod Update. 2010 May-Jun;16(3):231-45. doi: 10.1093/humupd/dmp048. Epub 2009 Nov 24. PMID 19934213
- [Background] Quintero RB, Urban R, Lathi RB, Westphal LM, Dahan MH. A comparison of letrozole to gonadotropins for ovulation induction, in subjects who failed to conceive with clomiphene citrate. Fertil Steril. 2007 Oct;88(4):879-85. doi: 10.1016/j.fertnstert.2006.11.166. PMID 17920403